CLINICAL TRIAL: NCT02198911
Title: The Effects of Chewing Gum on a Computer Task and Liking Ratings of Ice Cream
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 9212-B
Record Dates: First submitted 2014-03-25; First posted 2014-07-24 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Habituation
Keywords: Habituation; Orosensory cues; Satiation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Order 1 (Active Comparator): Gum chewing order for sessions, 1-3 respectively: NO GUM, MCC, C
  Interventions: Other: NO GUM; Other: MCC (Mint Chocolate Chip gum); Other: C (Cinnamon gum)
- Order 2 (Active Comparator): Gum chewing order for ice-cream sessions, 1-3 respectively: MCC, C, NO GUM
  Interventions: Other: NO GUM; Other: MCC (Mint Chocolate Chip gum); Other: C (Cinnamon gum)
- Order 3 (Active Comparator): Gum chewing order for ice-cream sessions, 1-3 respectively: C, NO GUM, MCC
  Interventions: Other: NO GUM; Other: MCC (Mint Chocolate Chip gum); Other: C (Cinnamon gum)

INTERVENTIONS:
Other: NO GUM — For the NO GUM condition, participants will not chew gum before engaging in a computer task that will allow participants to earn points for MCC ice cream that they can consume.
Other: MCC (Mint Chocolate Chip gum) — For the MCC gum condition, participants will chew MCC gum before engaging in a computer task that will allow participants to earn points for MCC ice cream that they can consume.
Other: C (Cinnamon gum) — For the C gum condition, participants will chew Cinnamon gum before engaging in a computer task that will allow participants to earn points for MCC ice cream that they can consume.

SUMMARY:
The purpose of this study is to examine if chewing gum before an eating bout will increase the rate of habituation and subsequently reduce energy intake within the eating bout.

DETAILED DESCRIPTION:
Approximately two-thirds of U.S. adults are overweight or obese, thus placing obesity first as a public health concern in the U.S. Not only is obesity detrimental at the individual level, by increasing risk for chronic disease and premature mortality, but it also presents problems at the economical level by increasing medical costs.

At the heart of weight management is the ability to appropriately regulate energy intake. A key factor in regulation of consumption is satiation, the process by which an eating bout ends. Quicker onset of satiation may result in decreased consumption, which is important in achieving an adequate energy balance. Negative energy balance, in which energy intake is less than energy expenditure, is required for weight loss; however, there are challenges with increased hunger and decreased satiation as energy intake is decreased.

One of the factors believed to influence satiation is the ability to increase the rate of habituation occurring during an eating bout. Habituation is a basic form of learning that can be measured by the rate of decrease in consummatory response to repeated presentations of food orosensory cues. Following this decreased response rate to a particular food, presentation of new orosensory cues may result in dishabituation to both the previously habituated food as well as the new orosensory cue, thus causing an increase in consummatory response. Dishabituation during an eating bout, i.e. exposure to a variety of orosensory cues, may be related to recovery of appetite and decreased satiation, leading the calorie-replete individual to overconsume. Alternatively, with repeated presentations of the same orosensory cue, one becomes accustomed to the taste faster, giving rise to habituation, which should increase satiation. A more rapid rate of habituation would mean that less energy is consumed within an eating bout. Research indicates increased weight status in relation to slower habituation rates as well as an inverse relationship between the extent of orosensory variety and habituation rates. Additionally, research shows a positive association between amount of orosensory cues and amount consumed within an eating bout.

One way to provide a single orosensory cue and initiate enhanced habituation with a minimal amount of additional energy intake is by chewing sugar-free, flavored gum. If matched to the flavor of the food about to be consumed, chewing gum prior to an eating bout may increase the rate of habituation, consequently reducing consumption.

Therefore, the purpose of this proof-of-concept study is to examine if chewing gum before an eating bout will increase the rate of habituation and subsequently reduce energy intake within the eating bout. The outcomes of this study may be useful in the health setting for creating prescriptions for weight-loss, weight maintenance, and weight-gain prevention.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* of normal weight (body mass index [BMI] between 18.5 and 24.9 kg/m2)
* unrestrained eater (scoring less than/equal to 12 on the restraint scale of the Three Factor Eating Questionnaire [TFEQ15])
* non-smoker (not having smoked or used tobacco products for a year or more)
* like and are willing to eat (greater than/equal to 50mm on a 100mm visual analogue scale [VAS]) MCC ice cream

Exclusion Criteria:

* have any health condition that requires a specific dietary prescription (i.e., diabetes)
* are unable to chew the gum for the time required in the investigation; 3) do not like the flavors of gum used in the investigation
* are allergic to any ingredients in the foods used in the investigation
* are lactose-intolerant
* plan to make any changes in dietary intake or physical activity over the course of the study
* score >20 on the Eating Attitudes Test (EAT8)
* score >16 on the Binge Eating Scale (BES10)
* are not able to stay within the metropolitan area within the time frame of the investigation
* are pregnant, lactating, or plan to become pregnant during the investigation
* are taking any type of medication that influences appetite.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grams of ice cream eaten | 3 trials (60 minutes)
  Amount of ice cream consumed will be measured using the following formula: amount of ice cream before consumption (first weight) - amount of ice cream following consumption (second weight). Grams of ice cream consumed will be determined following each 60 minute session (1, 2, and 3).

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Labroatory, University of Tennessee, Knoxville, Knoxville, Tennessee, United States